CLINICAL TRIAL: NCT00218894
Title: The Effect of Cataract Surgery on Gait, Balance and Falls in Older Persons
Brief Title: The Influence of Vision on Balance, Gait and Falls
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Midt-Norge (Other)
Responsible Party: Sponsor
Other Study IDs: 196-03; Helse Midt-Norge
Record Dates: First submitted 2005-09-20; First posted 2005-09-22 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cataract
Keywords: Effect; Balance; Gait; Falls
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- post cataract surgery
  Interventions: Procedure: Cataract surgery

INTERVENTIONS:
Procedure: Cataract surgery — surgery one one or two eyes by use of two different types of lenses and correcting for refraction

SUMMARY:
Falls are the most serious and frequent home accident amongst elderly. Most falls occur during walking. Vision is reduced with ageing and visual impairments affect balance. Uncorrected visual deficits and balance problems are reported to be risk factors for falls and fall related fractures. The present project uses a longitudinal design and aims at assessing the impact of cataract surgery on balance and gait as risk factors for falls.

DETAILED DESCRIPTION:
A longitudinal design is used, where subjects referred to the Cataract Unit are tested 1-3 weeks in advance of the surgery, and 4-6 weeks and 12 months after the surgery. Outcome measures are visual function, falls, balance and gait. Secondary outcome is quality of life, fear of falling and daily life functioning

ELIGIBILITY:
Inclusion Criteria:

* >70 years of age
* referred to cataract surgery on one or both eyes
* able to walk unassisted at least 10 m

Exclusion Criteria:

* terminal illness
* have undergone orthopedic surgery in the lower limbs the last 12 months
* Have had a stroke last 12 months
* dementia (measured by MMSE <20

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Elderly patients (70 years and older) referred to cataract surgery in StOlavs Hospital, Trondheim Norway.
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2004-01; Primary Completion 2008-03 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Falls | over one year
Visual function | pre surgery, 6-9 weeks and 1 year post surgery

SECONDARY OUTCOMES:
Health related Quality of Life | pre surgery, 6-9 weeks and one year after surgery
Gait | pre surgery, 6-9 weeks and one year after surgery
Fear of falling | pre surgery, 6-9 weeks and one year after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Olav Sletvold, Professor, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Section of Geriatric Medicine, St. Olavs University Hospital, Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Helbostad JL, Oedegaard M, Lamb SE, Delbaere K, Lord SR, Sletvold O. Change in vision, visual disability, and health after cataract surgery. Optom Vis Sci. 2013 Apr;90(4):392-9. doi: 10.1097/OPX.0b013e3182843f16. PMID 23422945